CLINICAL TRIAL: NCT05702697
Title: The Efficacy of Focus Extracorporeal Shock Wave Therapy on Hamstring Tightness in Healthy Subjects
Brief Title: The Efficacy of Focus Extracorporeal Shock Wave Therapy on Hamstring Tightness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Songsuda Roongsaiwatana, Principal Investigator, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COA. MURA2020/1084
Record Dates: First submitted 2023-01-06; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Hamstring Tightness

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F-ESWT (Experimental): F-EWST with 0.15 mJ/mm2 intensity and 6 Hz frequency for 3 weeks. The shocking head was placed at the muscle positions of the long head of the bicep femoris, semitendinosus, and semimembranosus for 1,000, 500, and 500 shocks, respectively, accounting for 2,000 shocks in total/ session/week.
  Interventions: Device: focus extracorporeal shock wave therapy; Behavioral: Home stretching program
- Sham-ESWT (Sham Comparator): sham ESWT by using the focused shockwave device and placing the shocking head in the same muscle positions as performed in the intervention group with 0.01 mJ/mm2 intensity and 6 Hz frequency in 2,000 shocks/session/week for 3 weeks.
  Interventions: Behavioral: Home stretching program

INTERVENTIONS:
Device: focus extracorporeal shock wave therapy — F-EWST with 0.15 mJ/mm2 intensity and 6 Hz frequency for 3 weeks. The shocking head was placed at the muscle positions of the long head of the bicep femoris, semitendinosus, and semimembranosus for 1,000, 500, and 500 shocks, respectively, accounting for 2,000 shocks in total/ session/week.
  Arms: F-ESWT
Behavioral: Home stretching program — The leaflet on hamstring stretching exercises (in a sitting posture)

SUMMARY:
To study efficacy of focus extracorporeal shock wave therapy on the flexibility of hamstring muscles in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Limited hamstring flexibility; passive knee extension degree >20
* No underlying disease

Exclusion Criteria:

* Patients with history of physical therapy in past 3 month
* Patient with analgesic drug such as muscle relaxant or NSAID.
* Patient with limited hamstring flexibility due to neurological or musculoskeletal diseases.
* Patient with cardiac pacemaker, pregnancy, hypercoagulable conditions, severe osteoporosis, malignancy or active infection around intervention site.
* Patient with history of chronic knee or back pain
* Patient cannot follow home stretching exercise program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Passive knee extension test | Immediately after every F-ESWT treatment, for 3sessions
  The clinician extends the knee until reaching the maximal tolerable stretch of the hamstring muscle as indicated by the patient with the ipsilateral hip remaining in 90 of flexion. The knee angle is then measured with a goniometer

SECONDARY OUTCOMES:
Back-saver sit-and-reach test (BSSR) | Immediately after every F-ESWT treatment, for 3sessions
Sit and reach test (SRT) | Immediately after every F-ESWT treatment, for 3sessions
Toe touch test (TT) | Immediately after every F-ESWT treatment, for 3sessions

CONTACTS AND LOCATIONS:
Overall Officials: Songsuda Roongsaiwatana, M.D., Study Director — Ramathibodi Hospital
Locations (1):
- Physical medicine and rehabilitation, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim YW, Chang WH, Kim NY, Kwon JB, Lee SC. Effect of Extracorporeal Shock Wave Therapy on Hamstring Tightness in Healthy Subjects: A Pilot Study. Yonsei Med J. 2017 May;58(3):644-649. doi: 10.3349/ymj.2017.58.3.644. PMID 28332373